CLINICAL TRIAL: NCT00499395
Title: Detection of Residual Colorectal Liver Metastases Within 24 Hours After RFA With 18-F FDG PET
Brief Title: Fludeoxyglucose F 18-PET Imaging for Early Detection of Residual Disease in Patients Undergoing Radiofrequency Ablation of Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 0513; CDR0000553137 (Other: PDQ number)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: positron emission tomography — All patients will undergo pre RFA PET prior to ablation for intra and extrahepatic staging and to assess FDG avidity of the lesions. When evaluating patients with liver metastases, we routinely obtain a dedicated liver PET study (Liver View) after the whole body PET. Patients will undergo two post RFA PET scans as part of this project: PET # 1) within 32 hours after RFA. The patients having percutaneous RFA will undergo PET on the same day after the clinical studies at the PET facility are completed; this will be within 8 hours after RFA. In case of laparoscopic and intra-operative RFA, PET will be performed on the following day after the clinical studies are completed; this will be within 32 hours after RFA. PET # 2) on day seven after RFA
Procedure: radiofrequency ablation — All patients will undergo pre RFA PET prior to ablation for intra and extrahepatic staging and to assess FDG avidity of the lesions. Patients will undergo two post RFA PET scans as part of this project: PET # 1) within 32 hours after RFA. The patients having percutaneous RFA will undergo PET on the same day after the clinical studies at the PET facility are completed; this will be within 8 hours after RFA. In case of laparoscopic and intra-operative RFA, PET will be performed on the following day after the clinical studies are completed; this will be within 32 hours after RFA. PET # 2) on day seven after RFA

SUMMARY:
RATIONALE: Diagnostic procedures, such as fludeoxyglucose F 18-PET imaging, may be effective in detecting residual disease after radiofrequency ablation of liver metastases in patients with colorectal cancer.

PURPOSE: This clinical trial is studying fludeoxyglucose F 18-PET imaging to see how well it works for early detection of residual disease in patients undergoing radiofrequency ablation of liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the sensitivity and specificity of fludeoxyglucose F 18 (FDG)-PET imaging in detecting residual disease within 48 hours after radiofrequency ablation (RFA) of liver metastases in patients with colorectal cancer.

Secondary

* Determine the findings on day 7 after RFA using FDG-PET imaging in these patients.

OUTLINE: This is a prospective study.

Patients undergo fludeoxyglucose F 18 (FDG)-PET imaging at baseline. They then undergo percutaneous laparoscopic or intraoperative radiofrequency ablation (RFA). Patients then undergo further FDG-PET scans within 48 hours and 7 days after RFA. FDG-PET images are evaluated for residual disease, including focal FDG uptake at the site of ablation. Beginning 1 month after RFA, patients undergo contrast-enhanced MRI for routine post-ablation follow-up. MRI scans are performed at 1, 4, 7, 12, 18, and 24 months after completion of RFA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer

  * Disease metastatic to the liver
* Undergoing percutaneous, intraoperative or laparoscopic radiofrequency ablation for liver metastases at the University of North Carolina Gastrointestinal Oncology Clinic

PATIENT CHARACTERISTICS:

* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No chemotherapy within 7 days after RFA on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of fludeoxyglucose F 18 (FDG)-PET imaging in early diagnosis of residual disease

SECONDARY OUTCOMES:
Findings on day 7 after RFA using FDG-PET imaging

CONTACTS AND LOCATIONS:
Overall Officials: Amir H. Khandani, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States